CLINICAL TRIAL: NCT05432479
Title: A Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy of a Probiotic in Infantile Colic Symptoms Relief
Brief Title: Study to Evaluate the Efficacy of a Probiotic in Infantile Colic Symptoms Relief
Acronym: PIXAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCTB202010
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Infantile Colic
Keywords: probiotic; Bifidobacterium; colic; cry
MeSH Terms: conditions — Colic; Crying | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Arm receiving investigation product (probiotic)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Arm receiving placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Single strain probiotic in a form of a sachets with a daily dose of 1.0E+9 Colony Forming Unit (CFU) per day for 4 weeks
  Arms: Active
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of single strain probiotic administered in a form of a sachet in the treatment of infant colic in infants 3-12 weeks old.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of minimum 37 weeks.
* Birthweight of minimum 2500 g (5.5 lb.).
* Age of greater than 3 weeks and less than 12 weeks at enrolment.
* Confirmed Infantile colic defined as: parental report of crying and/or fussing ≥3 hours/day for ≥3 days/week, confirmed prior to enrolment with an infant behaviour diary recording >3 hours of crying in a 24-hour period (eDiary App completed daily during run-in period & for duration of study).
* Participant Informed Consent form signed by parent or legal guardian.
* Infant is considered healthy following physical exam.
* Parents/Caregivers are willing to comply with the trial procedures, and the mother of the infant can attend all three trial visits

Exclusion Criteria:

* Use of antibiotics by the infant within 2-weeks prior to the screening visit or during the run-in period of the trial.
* Use of probiotic supplements from child's birth to enrolment (this includes infant formulas containing probiotics).
* Need for hospitalization (defined as readmission to a hospital ward after initial discharge following delivery).
* Congenital disorders that, in the opinion of the investigator, would impact the gastrointestinal tract.
* Failure to thrive.
* Known lactose or gluten intolerance.
* Known allergy to cow's milk proteins, fish, or any of the substances of the trial product or placebo.
* Known other causes for abdominal pain (e.g., pyloric stenosis).
* Participation in any other interventional clinical study.
* Immuno-compromised participant or participant with other severe chronic disorder.
* Use of probiotic supplements by breastfeeding mother from child's birth to enrolment.
* Use of antibiotics by breastfeeding mother within 2-weeks prior to the screening visit or during the run-in period of the trial.
* Any Participant/Parent/Caregiver who is an employee of the investigational site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in cry and fuss time | Day 0 , Day 28
  eDiary parent reported cry and fuss time

SECONDARY OUTCOMES:
Resolution of colic symptoms | Day 0, Day 28
  Reduction of cry and fuss time (parent reported) greater than 90% comparing to baseline
Change in cry and fuss time bouts | Day 0, Day 28
  eDiary parent reported cry and fuss bouts
Change in sleeping time | Day 0 Day 28
  eDiary parent reported sleep time
Change in the use of rescue medications | Day 0, Day 28
  Change in the proportion of participants needing to use rescue medications between the study arms

OTHER OUTCOMES:
Change in maternal quality of life and mental health | Day 0, Day 28
  Change in maternal QoL using WHO QOL/BREF (improvement marked by increase in the total score)
Change in maternal quality of life and mental health | Day 0, Day 28
  Change in maternal QoL using MMPP/QoL (improvement marked by increase in the total score)

CONTACTS AND LOCATIONS:
Locations (2):
- Atlantia Food Clinical Trials, Chicago, Illinois, United States
- Pulse Multispeciality Hospital,, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No